CLINICAL TRIAL: NCT04316923
Title: Analysis of Cardiac Biomarkers, Electrocardiograms and Cardio-pulmonary Exercise Test (CPET) Results in Children With Dilated (DCM), Hypertrophic (HCM) and Left-ventricle Non-compaction (LVNC) Cardiomyopathies
Brief Title: Analysis of Cardiac Biomarkers, ECG and CPET Results in Children With Cardiomyopathies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Katarzyna Łuczak-Woźniak (Other)
Responsible Party: Sponsor-Investigator, Katarzyna Łuczak-Woźniak, MD, Department of Pediatric Cardiology and General Pediatrics, Medical University of Warsaw, Warsaw, Poland., Medical University of Warsaw
Organization: Medical University of Warsaw (Other)
Other Study IDs: WUM CM
Record Dates: First submitted 2020-03-05; First posted 2020-03-20 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with cardiomyopathies: Children aged 0-18 years that have been diagnosed with DCM, HCM or LVNC on the basis of a two-dimensional echocardiography with color Doppler.
  Interventions: Diagnostic Test: ECG; Diagnostic Test: 24-hour ECG monitoring; Diagnostic Test: Cardio-pulmonary exercise test (CPET); Diagnostic Test: Cardiac biomarkers
- Healthy children: The control group will be composed of healthy children, in whom heart disease will be excluded using echocardiography.
  Interventions: Diagnostic Test: ECG; Diagnostic Test: 24-hour ECG monitoring; Diagnostic Test: Cardio-pulmonary exercise test (CPET)

INTERVENTIONS:
Diagnostic Test: ECG — ECG will be performed during each visit in the study group.
Diagnostic Test: 24-hour ECG monitoring — 24-hour ECG monitoring will be performed during each visit in the study group.
Diagnostic Test: Cardio-pulmonary exercise test (CPET) — CPET will be performed during the first and the last visit in the study group.
Diagnostic Test: Cardiac biomarkers — Cardiac biomarkers will be assessed during each visit in the study group.
  Groups: Children with cardiomyopathies

SUMMARY:
The aim of the study is to analyze cardiac biomarkers, electrocardiograms and cardio-pulmonary exercise test (CPET) results in children with cardiomyopathies.

DETAILED DESCRIPTION:
The study group will consist of children that have been diagnosed with DCM, HCM or LVNC. The control group will be composed of healthy children. Examination of cardiac biomarkers (in the study group), ECG, 24-hour- ECG monitoring, CPET will be performed.

Patients in the study group will be invited for 2 consecutive visits (in 6-10 months intervals). During the first and the last visit CPET will be performed. The control group will not be invited for consecutive visits.

ELIGIBILITY:
Inclusion Criteria:

* Children with HCM, DCM, LVNC diagnosed in 2D echo.
* Healthy children with no congenital heart disease (CHD) in 2D echo.
* Patients who signed consent form.

Exclusion Criteria:

* Patients with coexisting CHD, kidney and liver disfunction, taking anti-psychotic and anti-depressant medication, or patients with bundle bunch blocks in ECG.
* no consent form signed.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study group will consist of children aged 0-18 years that have been diagnosed with DCM, HCM or LVNC who are under the care of our Deparment.
  The control group will be composed of 30 healthy children, in whom heart disease will be excluded using echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Assessment of ECG (electrocardiographic) differences in children with cardiomyopathies and healthy children. | 14 months
  Assessment of heart rhythm, heart rate (BPM), PQ, QRS, QT, QTc intervals, QRS-T angle and arrythmia in ECG. These will be compared with arrythmia severity in 24-hour ecg monitoring.
Assessment of differences in CPET results in children with cardiomyopathies and healthy children. | 14 months
  Assessment of peak respiratory oxygen uptake (peakVo2), carbon dioxide production (Vco2), anaerobic threshold (AT), expired ventilation (VE), ventilatory equivalent for CO2 (VE/VCO2), VO2/Work rate relationship, maximal workload (W), duration of exercise (T).

SECONDARY OUTCOMES:
Assessment of progression of heart failure in children with cardiomyopathies | 20 months
  Assessment of serum cardiac biomarkers (Troponin I, NT-proBNP) in children with cardiomyopathies during each visit.
Assessment of arrhythmia in time in children with cardiomyopathies | 20 months
  Assessment of heart rhythm, heart rate (BPM), PQ, QRS, QT, QTc intervals, QRS-T angle and arrythmia in ECG during each control visit. The results will be compared to the severity of arrythmia in 24-hour ecg monitoring. These test will be performed during each visit.
Assessment of changes in CPET results in children with cardiomyopathies | 20 months
  Assessment of peak respiratory oxygen uptake (peakVo2), carbon dioxide production (Vco2), anaerobic threshold (AT), expired ventilation (VE), ventilatory equivalent for CO2 (VE/VCO2), VO2/Work rate relationship, maximal workload (W), duration of exercise (T). CPET will be performed in during the first and the last control visit.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna M Luczak-Wozniak, MD, Principal Investigator — Medical Univeristy of Warsaw, Poland
Locations (1):
- Medical Univeristy of Warsaw, Warsaw, Poland